CLINICAL TRIAL: NCT02866903
Title: IPOXA, Phase I/II Dose Escalation Trial Aiming to Evaluate the Safety of Intraperitoneal (IP) OXAliplatin (OXA) in Association With Systemic FOLFIRI Bevacizumab Chemotherapy in Patients With Peritoneal Carcinosis of Colorectal Origin and Uncertain Resectability.
Brief Title: Safety of Intraperitoneal (IP) OXAliplatin (OXA) in Association With Systemic FOLFIRI Bevacizumab Chemotherapy in Patients With Peritoneal Carcinosis
Acronym: IPOXA
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 69HCL16_0134
Record Dates: First submitted 2016-08-04; First posted 2016-08-15 (Estimated); Last update posted 2017-09-21 (Actual); Status verified 2017-09

CONDITIONS: Peritoneal Carcinosis
Keywords: Peritoneal carcinosis; intraperitoneal (IP) OXAliplatin; Phase I/II dose escalation trial; FOLFIRI Bevacizumab chemotherapy
MeSH Terms: interventions — Infusions, Parenteral; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with peritoneal carcinosis (Experimental): Patients with peritoneal carcinosis of colorectal origin and uncertain resectability with an indication for systemic chemotherapy compatible with the FOLFIRI + bevacizumab combination.
  Interventions: Drug: intraperitoneal (IP) OXAliplatin (OXA) + systemic FOLFIRI bevacizumab chemotherapy

INTERVENTIONS:
Drug: intraperitoneal (IP) OXAliplatin (OXA) + systemic FOLFIRI bevacizumab chemotherapy — Intraperitoneal (IP) OXAliplatin (OXA) in association with systemic FOLFIRI bevacizumab chemotherapy Intraperitoneal (IP) OXAliplatin (OXA) + systemic FOLFIRI (Irinotecan IV + 5-FU IV) bevacizumab chemotherapy in escalation dose (every 14 days) starting with the level 1
Drug: intraperitoneal (IP) OXAliplatin (OXA) + systemic FOLFIRI bevacizumab chemotherapy — systemic FOLFIRI chemotherapy
Drug: intraperitoneal (IP) OXAliplatin (OXA) + systemic FOLFIRI bevacizumab chemotherapy — bevacizumab

SUMMARY:
Peritoneal carcinosis (PC) corresponds to a locoregional extension into the peritoneum of rare primary peritoneal cancers, or more frequently distant extension of digestive cancers (colorectal or gastric) or gynecological (ovarian, fallopian tube, or endometrial). PC can be considered as a distinct oncological entity as its genesis, natural history, and response to systematic treatments differ to those of other metastases. The development of PC, observed in 25-35% of colorectal cancers, is generally considered as a unfavorable event in the course of the disease. The prognosis is defined by the possibility of complete resection, possibly after neoadjuvant treatment. The benefit provided by the combination of cytoreductive surgery and heated intraperitoneal chemotherapy (HIPEC) with respect to systemic chemotherapy in patients with PC of colorectal origin has been demonstrated based on overall survival in several randomized trials, among which one evaluated oxaliplatin. The evaluation of the clinical benefit-risk related to the repeated administration of non-hyperthermic intraperitoneal chemotherapy, as has been validated in ovarian cancer, in patients with PC of colorectal origin is already being investigated by several international teams.

The FOLFOXIRI + bevacizumab every 2 weeks is a modern therapeutic option in patients with this disease. The intraperitoneal rather than intravenous (IV) administration of oxaliplatin, in this combination, could increase the response of peritoneal lesions known to be relatively insensitive to IV chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old and ≤ 75 years old
* ECOG Performance Status (PS) 0-2
* Peritoneal carcinosis with locoregional extension or metastases of colorectal origin and uncertain resectability
* PCI > 20 and / or infiltration of the hepatic pedicle and / or necessary digestive tract resections
* Systemic chemotherapy indication, compatible with the FOLFIRI + bevacizumab combination
* Satisfactory haematological evaluation: PNN rate greater than 1500 / mm3, platelet count greater than 100 G / l;
* Satisfactory renal and hepatic function : serum creatinine ≤1.5 times the normal lower values or creatinine clearance ≥50 ml / min, bilirubin ≤1.25 times lower normal values, AST / ALT ≤1.5 times the lower normal values (≤5 times the lower normal values for patients with liver metastases)
* No unstable conditions: myocardial infarction within 6 months prior to the start of the study, congestive heart failure, unstable angina, active cardiomyopathy, unstable rhythm disorder, uncontrolled hypertension, uncontrolled psychiatric disorders, severe infection, peptic ulcer or any condition that could be aggravated by treatment or limit compliance (investigator assessment);
* No limitation in the number of previous treatments;
* Patients may have received conventional cytotoxic chemotherapy , hormonal or immunological targeted biological agents. They should have recovered from previous grade ≤2 toxicities
* Written informed consent
* Known RAS status.

Exclusion Criteria:

* Extraperitoneal metastases for which the site or number preclude potentially curative surgery at any moment during the course of the disease
* Sign of bowel obstruction or lesions whose topography indicates a risk of intestinal perforation or inflammatory bowel disease
* ECOG PS 3-4
* Contraindication to the placement of a intraperitoneal central line
* Contraindication specifically related to intraperitoneal administration of oxaliplatin
* known history of hypersensitivity to oxaliplatin or to the excipients
* peripheral sensory neuropathy grade ≥2
* Pregnant or lactating women
* Unable to give consent
* Patient under legal protection measures
* Refusal to participate in the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Estimated)
Dates: Start 2017-05-18 (Actual); Primary Completion 2019-03 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
Adverse events (NCI CTCAE v4.0) | up to 14 days
  The safety of intraperitoneal (IP) administration of oxaliplatin in combination with systemic chemotherapy FOLFIRI + bevacizumab will be evaluated during the first cycle of therapy according to NCI CTCAE version 4.0
Dose Limiting Toxicities, DLT | up to 14 days
  The safety of intraperitoneal (IP) administration of oxaliplatin in combination with systemic chemotherapy FOLFIRI + bevacizumab will be evaluated during the first cycle of therapy according to Dose Limiting Toxicities

SECONDARY OUTCOMES:
Overall response rate according to RECIST | up to 4 months
  Clinical efficacy of intraperitoneal (IP) administration of oxaliplatin in combination with systemic FOLFIRI + bevacizumab assessed by the overall response rate according to RECIST version 1.1 criteria assessed by imaging (TAP scanner and / or MRI if contraindication) performed after 4 cycles, and / or after 8 cycles
Peritoneal Cancer Index (PCI) | up to 4 months
  Clinical efficacy of intraperitoneal (IP) administration of oxaliplatin in combination with systemic FOLFIRI + bevacizumab assessed by Peritoneal Cancer Index (PCI) performed after 4 cycles, and / or after 8 cycles
Adverse events (NCI CTCAE v4.0) | up to 5 months
  The safety of intraperitoneal (IP) administration of oxaliplatin in combination with systemic chemotherapy FOLFIRI + bevacizumab will be evaluated throughout the duration of treatment (4 months) and until the end of patient follow up (1 month after treatment discontinuation) according to NCI CTCAE version 4.0
The quality of life (EORTC QLQ-C30) | up to 4 months
  The quality of life will be evaluated throughout the duration of treatment (4 months max) after the end of cycle 2, 4, 6 and 8 of chemotherapy according to EORTC QLQ-C30 .
The quality of life (EORTC QLQ-C29) | up to 4 months
  The quality of life will be evaluated throughout the duration of treatment (4 months max) after the end of cycle 2, 4, 6 and 8 of chemotherapy according to EORTC QLQ-C29.

CONTACTS AND LOCATIONS:
Overall Officials: Benoit You, MD, Principal Investigator — Service d'Oncologie Médicale, Hospices Civils de Lyon, Centre Hospitalier Lyon Sud 69495 Pierre-Bénite
Locations (6):
- France (6):
  - CHU Estaing, Clermont-Ferrand
  - Service de Chirurgie Digestive et de l'Urgence, CHU Albert Michallon, Grenoble
  - Département de Chirurgie Cancérologique, Centre Léon Bérard, Lyon
  - Service d'Oncologie Médicale, Hospices Civils de Lyon, Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Service de Chirurgie Digestive et Cancérologique, CHU NORD, Saint-Etienne
  - Service Oncologie Médicale, INSTITUT DE CANCEROLOGIE DE LA LOIRE (ICL), Saint-Priest-en-Jarez